CLINICAL TRIAL: NCT02917174
Title: National Mobile Asthma Management System-E Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jiangtao Lin, Chief physician, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CARN2016-01
Record Dates: First submitted 2016-08-08; First posted 2016-09-28 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Asthma
Keywords: asthma; m-health; asthma control; self-management
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobile management (Experimental): use mobile management to improve asthma control
  Interventions: Behavioral: Mobile Asthma Management System
- Traditional management (Other): use Traditional management to improve asthma control
  Interventions: Behavioral: traditional Asthma Management System

INTERVENTIONS:
Behavioral: Mobile Asthma Management System — Patients in this group use a smartphone app in their asthma self-management.
  Arms: mobile management
Behavioral: traditional Asthma Management System — Patients in this group use a printed asthma diary in their asthma self-management.
  Arms: Traditional management

SUMMARY:
Bronchial asthma is a heterogeneous disease characterized by chronic airway inflammation, which is a common and frequently occurring disease in the world, and has resulted in a sustained increase of social and economic burden. However, several studies suggest, lots of asthma patients did not get their asthma controlled. The investigators study showed that in China only 28.7% of asthma patients achieve asthma controlled during 2007-2008. In recent years, application softwares of mobile-phones for asthma have gradually increased, studies suggested that application of these application softwares can make treatment more standard, reduce asthma attacks, help patients to control their asthma, improve adherence and these application softwares also show many other advantages. This study is a prospective, multi center, randomized, controlled study, aims to evaluate the efficacy of application softwares in asthma patients, provide a new tool to asthma management.

ELIGIBILITY:
Inclusion Criteria:

1.18 years of age or older, having been resided in the same city during the study; 2.A history of at least 3 months of diagnosed asthma based on the criteria established by GINA 2016; need to be on medication containing ICS or ICS/LABA 3.Asthma out patients with ACT scores﹤20 and MARS - A mean score < 4.5 ; 4.Owning and Being able to use smart phone that the corresponding software can be successfully installed; 5.Subjects who are willing to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Unable to communicate properly because of visual impairment, hearing impairment and language barrier, or with mental illness or psychological problems;
2. Have a history of tracheal intubation or mechanical ventilation as a result of acute asthma attack;
3. Have respiratory tract infection within the prior 4 weeks; history of thoracic surgery; with comorbidities such as other/structural lung diseases (COPD, bronchiectasis, lung cancer, et al); heart disease; kidney or autoimmunity disease; or other conditions that could potentially effect asthma control or asthma disease status by investigator's medical opinion.
4. Women with pregnancy, or planned pregnancy within one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 870 (Actual)
Dates: Start 2017-03-25 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Proportion of good adherence at the 6th month | 6 months
  patients will fill out the MARS-A questionnaire on their own，and the MARS-A Scores will be calculated to show their adherence of medication. Good adherence: MARS-A score>=4.5

SECONDARY OUTCOMES:
Forced expiratory volume in one second（FEV1） | 1 year
  patients will accomplish the pulmonary function test，and the percentage of actual value to predicted value of FEV1 will be calculated to show their pulmonary function.(The predicted value of FEV1 can be calculated when age,gender,height and weight are already known.)
Forced vital capacity(FVC) | 1 year
  patients will accomplish the pulmonary function test，and the percentage of actual value to predicted value of FVC will be calculated to show their pulmonary function.
Peak expiratory flow(PEF) | 1 year
  patients will accomplish the pulmonary function test，and the percentage of actual value to predicted value of PEF will be calculated to show their pulmonary function.
Emergency visits | 1 year
  patients will report their times of emergency visits to the researchers.
Hospitalization | 1 year
  patients will report their times of hospitalization to the researchers.
Asthma Control Test（ACT） | 1 year
  patients will fill out the ACT questionnaire on their own，and the ACT Scores of 25 is classified as well-controlled asthma，between 20 and 24 as not well-controlled，and less than 20 as poorly controlled asthma. ACT score is used to describe the proportion of people with different levels of asthma control.
Proportion of good adherence | 1 year
  patients will fill out the MARS-A questionnaire on their own，and the MARS-A Scores will be calculated to show their adherence of medication. Good adherence: MARS-A score>=4.5. Compare the proportion of good adherence change with time, time points: 1st month, 2nd month, 3rd month, 6th month, 12th month.
Asthma Quality of Life Questionnaire(AQLQ) | 1 year
  patients will fill out the AQLQ questionnaire on their own，and the AQLQ Scores will be calculated to show their quality of life.
Correct answer rate of the given asthma awareness questions | 1 year
  patients will answer 4 questions about asthma, correct answer rate will be calculated to show their awareness of asthma.
Fractional exhaled nitric oxide(FeNO) | 1year
  patients will accomplish the fractional exhaled nitric oxide test，and the result of fractional exhaled nitric oxide related to airway inflammation.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Lin J, Wang W, Tang H, Huo J, Gu Y, Liu R, Chen P, Yuan Y, Yang X, Xu J, Sun D, Li N, Jiang S, Chen Y, Wang C, Yang L, Liu X, Yang D, Zhang W, Chen Z, Lin Q, Liu C, Zhou J, Zhou X, Hu C, Jiang P, Zhou W, Zhang J, Cai S, Qiu C, Huang M, Huang Y, Liu H; China Asthma Research Collaboration Network. Asthma Management Using the Mobile Asthma Evaluation and Management System in China. Allergy Asthma Immunol Res. 2022 Jan;14(1):85-98. doi: 10.4168/aair.2022.14.1.85. PMID 34983109